CLINICAL TRIAL: NCT06504862
Title: The Effect of Zongertinib on the Pharmacokinetics of Dabigatran (Part 1) and Rosuvastatin, Metformin and Furosemide Administered as a Cocktail (Part 2) in Healthy Male Subjects (a 2-part, Open-label, 2-period, Fixed-sequence Cross-over Trial)
Brief Title: A Study in Healthy Men to Test Whether Zongertinib Influences the Amount of 4 Other Medicines (Dabigatran, Rosuvastatin, Metformin, and Furosemide) in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0015; 2024-510628-38-00 (Registry Identifier: CTIS); U1111-1302-1171 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Rosuvastatin Calcium; Metformin; Furosemide

STUDY DESIGN:
Intervention Model Description: fixed-sequence crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: dabigatran-etexilate (R), then zongertinib and dabigatran-etexilate (T) (Experimental): Participants were administered a 150 milligram (mg) dabigatran-etexilate hard capsule orally with 240 milliliters (mL) of water after an overnight fast of at least 10 hours on Day 1 of period 1 (Reference treatment, R). After a wash-out period, participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally, and a 150 mg dabigatran-etexilate hard capsule orally on Day 1 of period 2 (Test treatment, T). Both medications were administered with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: Zongertinib; Drug: Dabigatran-etexilate
- Part 2: drug cocktail (R), then zongertinib and drug cocktail (T) (Experimental): Participants were administered a cocktail consisting of a 10 mg rosuvastatin film-coated tablet, a 10 mg metformin oral solution, and a 1 mg furosemide oral solution with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of period 1 (Reference treatment, R). In period 2, from Day -9 to Day 3, participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally every day. On Day 1, participants were also administered a cocktail consisting of a 10 mg rosuvastatin film-coated tablet, a 10 mg metformin oral solution, and a 1 mg furosemide oral solution (Test treatment, T). Every medication was administered with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: Zongertinib; Drug: Rosuvastatin; Drug: Metformin hydrochloride; Drug: Furosemide

INTERVENTIONS:
Drug: Zongertinib — A 120 mg dose on Day 1 of period 2 (Part 1) OR daily (Part 2) with 240 mL of water after an overnight fast of at least 10 hours.
  Other Names: Hernexeos®
Drug: Dabigatran-etexilate — A 150 mg dose on Day 1 of each period with 240 mL of water after an overnight fast of at least 10 hours.
  Other Names: Pradaxa®
  Arms: Part 1: dabigatran-etexilate (R), then zongertinib and dabigatran-etexilate (T)
Drug: Rosuvastatin — A 10 mg dose on Day 1 of each period with 240 mL of water after an overnight fast of at least 10 hours.
  Other Names: Crestor®
  Arms: Part 2: drug cocktail (R), then zongertinib and drug cocktail (T)
Drug: Metformin hydrochloride — A 10 mg dose on Day 1 of each period with 240 mL of water after an overnight fast of at least 10 hours.
  Other Names: MetfoLiquid GeriaSan®
  Arms: Part 2: drug cocktail (R), then zongertinib and drug cocktail (T)
Drug: Furosemide — A 1 mg dose on Day 1 of each period with 240 mL of water after an overnight fast of at least 10 hours.
  Other Names: Lasix®
  Arms: Part 2: drug cocktail (R), then zongertinib and drug cocktail (T)

SUMMARY:
For Part 1 of the trial, the main objective is to assess the effect of a single dose of zongertinib on the pharmacokinetics of a single dose of dabigatran-etexilate. For Part 2 of the trial, the main objective is to assess the effect of zongertinib at steady-state on the pharmacokinetics of a single dose of rosuvastatin, metformin and furosemide (administered as a cocktail).

ELIGIBILITY:
Inclusion Criteria :

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria :

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomised, open-label, 2-period fixed-sequence crossover trial in healthy male participants to compare the test treatments (T: zongertinib and dabigatran-etexilate in part 1; zongertinib, rosuvastatin, metformin, furosemide in part 2) to the reference treatments (R: dabigatran-etexilate in part 1; rosuvastatin, metformin, furosemide in part 2).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not included in the trial if any of the entry criteria were violated.
Period: Period 1, reference treatment (R)
Arm/Group | Part 1: Dabigatran-etexilate (R), Then Zongertinib and Dabigatran-etexilate (T) | Part 2: Drug Cocktail (R), Then Zongertinib and Drug Cocktail (T)
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Transition period
Arm/Group | Part 1: Dabigatran-etexilate (R), Then Zongertinib and Dabigatran-etexilate (T) | Part 2: Drug Cocktail (R), Then Zongertinib and Drug Cocktail (T)
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2, test treatment (T)
Arm/Group | Part 1: Dabigatran-etexilate (R), Then Zongertinib and Dabigatran-etexilate (T) | Part 2: Drug Cocktail (R), Then Zongertinib and Drug Cocktail (T)
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all participants who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dabigatran-etexilate (R), Then Zongertinib and Dabigatran-etexilate (T) | Part 2: Drug Cocktail (R), Then Zongertinib and Drug Cocktail (T) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (9.4) | 37.8 (11.2) | 36.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve of Dabigatran in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of dabigatran in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: Within 3 hours (h) before dabigatran-etexilate administration (R only), within 3 h prior to zongertinib administration (T only), and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 34, 48 h after dabigatran-etexilate administration (R and T).
Population: Pharmacokinetic parameter analysis set (PKS) restricted to part 1: all part 1 participants in the TS who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a participant was included in the PKS, even if he contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanogram/milliliter (h*ng/mL)
Groups:
- Dabigatran-etexilate (R): Participants were administered a 150 mg dabigatran-etexilate hard capsule orally with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of period 1 (Reference treatment, R).
- Zongertinib and dabigatran-etexilate (T): Participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally, and a 150 mg dabigatran-etexilate hard capsule orally on Day 1 of period 2 (Test treatment, T). Both medications were administered with 240 mL of water after an overnight fast of at least 10 hours.
Arm/Group | Dabigatran-etexilate (R) | Zongertinib and dabigatran-etexilate (T)
Number analyzed (Participants) | 16 | 15
hour*nanogram/milliliter (h*ng/mL) | 725.25 (NA) — Adjusted geometric standard error = 1.12 | 971.67 (NA) — Adjusted geometric standard error = 1.12
Statistical Analysis 1: Comparison: Dabigatran-etexilate (R) vs Zongertinib and dabigatran-etexilate (T); Ratio of adjusted geometric means was calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale; Test type: Other; Ratio of adjusted geometric means [%] = 133.98, 90% CI 2-sided [105.52 to 170.11], Standard Error of Mean 1.15 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 39.0

2. Primary Outcome: Part 1: Maximum Measured Concentration of Dabigatran in Plasma (Cmax)
Description: Maximum measured concentration of dabigatran in plasma (Cmax) is reported. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanogram/milliliter (ng/mL)
Arm/Group | Dabigatran-etexilate (R) | Zongertinib and dabigatran-etexilate (T)
Number analyzed (Participants) | 16 | 15
nanogram/milliliter (ng/mL) | 89.01 (NA) — Adjusted geometric standard error = 1.13 | 110.53 (NA) — Adjusted geometric standard error = 1.13
Statistical Analysis 1: Comparison: Dabigatran-etexilate (R) vs Zongertinib and dabigatran-etexilate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 124.19, 90% CI 2-sided [96.13 to 160.43], Standard Error of Mean 1.16 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 42.0

3. Primary Outcome: Part 2: Area Under the Concentration-time Curve of Rosuvastatin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: Within 3 h prior to drug cocktail administration (R), within 15 minutes prior to drug cocktail and zongertinib administration (T), and 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 h after drug cocktail administration (R and T).
Population: Pharmacokinetic parameter analysis set (PKS) restricted to part 2: all part 2 participants in the TS who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a participant was included in the PKS, even if he contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Groups:
- Drug cocktail (R): Participants were administered a cocktail consisting of a 10 mg rosuvastatin film-coated tablet, a 10 mg metformin oral solution, and a 1 mg furosemide oral solution with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of period 1 (Reference treatment, R).
- Zongertinib and drug cocktail (T): In period 2, from Day -9 to Day 3, participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally every day. On Day 1, participants were also administered a cocktail consisting of a 10 mg rosuvastatin film-coated tablet, a 10 mg metformin oral solution, and a 1 mg furosemide oral solution (Test treatment, T). Every medication was administered with 240 mL of water after an overnight fast of at least 10 hours.
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
hour*nanomole/liter (h*nmol/L) | 102.98 (NA) — Adjusted geometric standard error = 1.10 | 237.15 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 230.30, 90% CI 2-sided [195.68 to 271.04], Standard Error of Mean 1.10 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 26.7

4. Primary Outcome: Part 2: Maximum Measured Concentration of Rosuvastatin in Plasma (Cmax)
Description: Maximum measured concentration of rosuvastatin in plasma (Cmax) is reported. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liter (nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
nanomole/liter (nmol/L) | 8.87 (NA) — Adjusted geometric standard error = 1.12 | 26.75 (NA) — Adjusted geometric standard error = 1.12
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 301.68, 90% CI 2-sided [247.19 to 368.19], Standard Error of Mean 1.12 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 33.0

5. Primary Outcome: Part 2: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
hour*nanomole/liter (h*nmol/L) | 1355.69 (NA) — Adjusted geometric standard error = 1.04 | 1125.52 (NA) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 83.02, 90% CI 2-sided [76.48 to 90.12], Standard Error of Mean 1.05 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 13.3

6. Primary Outcome: Part 2: Maximum Measured Concentration of Metforminin in Plasma (Cmax)
Description: Maximum measured concentration of metforminin in plasma (Cmax) is reported. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liter (nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
nanomole/liter (nmol/L) | 230.25 (NA) — Adjusted geometric standard error = 1.06 | 174.00 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 75.57, 90% CI 2-sided [68.03 to 83.95], Standard Error of Mean 1.06 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 17.1

7. Primary Outcome: Part 2: Area Under the Concentration-time Curve of Furosemide in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of furosemide in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
hour*nanomole/liter (h*nmol/L) | 172.84 (NA) — Adjusted geometric standard error = 1.07 | 238.43 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 137.95, 90% CI 2-sided [120.17 to 158.36], Standard Error of Mean 1.08 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 22.5

8. Primary Outcome: Part 2: Maximum Measured Concentration of Furosemide in Plasma (Cmax)
Description: Maximum measured concentration of furosemide in plasma (Cmax) is reported. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/liter (nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
nanomole/liter (nmol/L) | 75.73 (NA) — Adjusted geometric standard error = 1.11 | 113.45 (NA) — Adjusted geometric standard error = 1.11
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 149.80, 90% CI 2-sided [116.12 to 193.25], Standard Error of Mean 1.16 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 44.4

9. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of Dabigatran in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of dabigatran in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Dabigatran-etexilate (R) | Zongertinib and dabigatran-etexilate (T)
Number analyzed (Participants) | 16 | 15
hour*nanogram/milliliter (h*ng/mL) | 700.45 (NA) — Adjusted geometric standard error = 1.12 | 942.02 (NA) — Adjusted geometric standard error = 1.13
Statistical Analysis 1: Comparison: Dabigatran-etexilate (R) vs Zongertinib and dabigatran-etexilate (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 134.49, 90% CI 2-sided [105.56 to 171.34], Standard Error of Mean 1.15 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 39.5

10. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of Rosuvastatin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of rosuvastatin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
hour*nanomole/liter (h*nmol/L) | 93.10 (NA) — Adjusted geometric standard error = 1.10 | 231.53 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 248.69, 90% CI 2-sided [211.03 to 293.07], Standard Error of Mean 1.10 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 27.0

11. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
hour*nanomole/liter (h*nmol/L) | 1343.93 (NA) — Adjusted geometric standard error = 1.04 | 1113.21 (NA) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 82.83, 90% CI 2-sided [76.27 to 89.96], Standard Error of Mean 1.05 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 13.4

12. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of Furosemide in in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of furosemide in in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an ANOVA model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: participant (considered as random) and treatment (considered as fixed). These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | Drug cocktail (R) | Zongertinib and drug cocktail (T)
Number analyzed (Participants) | 16 | 16
hour*nanomole/liter (h*nmol/L) | 164.01 (NA) — Adjusted geometric standard error = 1.07 | 235.33 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: Drug cocktail (R) vs Zongertinib and drug cocktail (T); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 143.49, 90% CI 2-sided [123.78 to 166.33], Standard Error of Mean 1.09 — Ratio [%] = (adjusted geometric mean T/adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 24.2

ADVERSE EVENTS:
Time Frame: All adverse events occurring after 1st drug administration within treatment-specific time frames after end of administration, OR until next treatment administration, were assigned to treatment. The time frames for each treatment are: 3 days (dabigatran-etexilate), 6 days (cocktail), 14 days (zongertinib, zongertinib and dabigatran-etexilate, zongertinib and cocktail). All-cause mortality time frame: from drug administration until end of study, up to 30 days.
Description: Treated set (TS): all participants who were treated with at least one dose of trial drug.
Groups:
- Part 1: Dabigatran-etexilate (R): Participants were administered a 150 mg dabigatran-etexilate hard capsule orally with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of period 1 (Reference treatment, R).
- Part 1: Zongertinib: Participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of period 2.
- Part 1: Zongertinib and Dabigatran-etexilate (T): On Day 1 of period 2, after zongertinib administration, participants were administered a 150 mg dabigatran-etexilate hard capsule orally with 240 mL of water after an overnight fast of at least 10 hours (Test treatment, T).
- Part 2: Drug Cocktail (R): Participants were administered a cocktail consisting of a 10 mg rosuvastatin film-coated tablet, a 10 mg metformin oral solution, and a 1 mg furosemide oral solution with 240 mL of water after an overnight fast of at least 10 hours on Day 1 of period 1 (Reference treatment, R).
- Part 2: Zongertinib: In period 2, from Day -9 to Day -1, participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally every day.
- Part 2: Zongertinib and Drug Cocktail (T): Participants were administered a cocktail consisting of a 10 mg rosuvastatin film-coated tablet, a 10 mg metformin oral solution, and a 1 mg furosemide oral solution on Day 1 of period 2. On the same day, and up to Day 3, participants were administered two 60 mg film-coated tablets of zongertinib (total dose: 120 mg) orally every day (Test treatment, T).
Arm/Group | Part 1: Dabigatran-etexilate (R) | Part 1: Zongertinib | Part 1: Zongertinib and Dabigatran-etexilate (T) | Part 2: Drug Cocktail (R) | Part 2: Zongertinib | Part 2: Zongertinib and Drug Cocktail (T)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 0/15 | 3/15 | 5/16 | 9/16 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dabigatran-etexilate (R) (N=16) | Part 1: Zongertinib (N=15) | Part 1: Zongertinib and Dabigatran-etexilate (T) (N=15) | Part 2: Drug Cocktail (R) (N=16) | Part 2: Zongertinib (N=16) | Part 2: Zongertinib and Drug Cocktail (T) (N=16)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT06504862/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT06504862/SAP_001.pdf